CLINICAL TRIAL: NCT03370536
Title: Panoramic ECGi to Guide Ablation of Non-Paroxysmal AF: Effect of Ibutilide on AF Source Location and Organization
Brief Title: ECGi Ibutilide: Effect of Ibutilide on AF Source Location and Organization
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 1 patient enrolled (consented) but screen failed. Study stopped as unable to enroll.
Sponsor: Vivek Reddy (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor-Investigator, Vivek Reddy, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 40-5004
Record Dates: First submitted 2017-12-04; First posted 2017-12-12 (Actual); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-01

CONDITIONS: Atrial Fibrillation; Persistent Atrial Fibrillation
Keywords: Atrial Fibrillation; Persistent Atrial Fibrillation; AFIB; Arrhythmia
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac | interventions — ibutilide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Patients with AF (Experimental): Patients with AF and planned to undergo first catheter procedure
  Interventions: Device: CardioInsight ECGI Mapping System; Procedure: AF ablation; Drug: Ibutilide

INTERVENTIONS:
Device: CardioInsight ECGI Mapping System — The CardioInsight mapping system is a noninvasive, single beat cardiac arrhythmia mapping system that provides 3D electroanatomic maps of the heart.
  Other Names: ECGi mapping
Procedure: AF ablation — Empiric ablation (CFAE or linear ablation) is not permitted
  Other Names: Biosense Thermocool SF; Biosense Smart Touch SF (STSF)
Drug: Ibutilide — Progressive doses of Ibutilide administered (0.25mg, then 0.25mg, then 0.5mg)

SUMMARY:
This is a prospective, multi-center, non-randomized, un-blinded, observational trial.

DETAILED DESCRIPTION:
This prospective, multicenter observational study will examine the ability of ECGi mapping to

1. Effect of Ibutilide on the number and size of the driver domains
2. Effect of ablation of Ibutilide-organized driver domains
3. Effect of PV isolation on driver domains

The researchers hypothesize that this approach will lead to successful arrhythmia control .

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age.
* ° Symptomatic persistent AF refractory or intolerant to at least 1 class I or III antiarrhythmic medication Persistent AF - defined as Persistent: AF that is sustained > 7 days. Episodes of AF which are terminated by electrical or pharmacologic cardioversion after ≥ 48 hours of AF, but prior to 7 days, should also be classified as persistent AF episodes.

  * Planned to undergo first catheter ablation procedure ( prior atrial flutter typical is allowed)
* Ability to understand the requirements of the study and sign the informed consent form.
* Willingness to adhere to study restrictions and comply with all post-procedural follow-up requirements
* Projected lifespan greater than 1 year

Exclusion Criteria:

* They have baseline prolonged QT or renal failure precluding safe used of ibutilide
* Rheumatic heart disease,
* Current intra-cardiac thrombus,
* History of MI or CABG within 6 weeks;
* Class IV HF,
* Unable to sign consent
* Projected lifespan of < 1 year
* Women known to be pregnant or to have positive beta-HCG.
* Participation in another study that would interfere with this study.
* Unstable Angina
* Recent cerebral ischemic events
* Contraindication to anticoagulation
* Prior history of polymorphic ventricular tachycardia or torsades de pointes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Koruth, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Vivek Reddy, MD, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With AF
Started | 1
Completed | 0
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Patients With Atrial Fibrillation (AF): Patients with AF and planned to undergo first catheter procedure
Arm/Group | Patients With Atrial Fibrillation (AF)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who no Longer Has Recurrent At/AF
Description: Freedom from recurrent At/AF
Time Frame: at 12 months
Population: Participant screen failed
Arm/Group | Patients With Atrial Fibrillation (AF)
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Drivers
Description: Number of drivers identified
Time Frame: Baseline
Population: Participant screen failed
Arm/Group | Patients With Atrial Fibrillation (AF)
Number analyzed (Participants) | 0

3. Secondary Outcome: Size of Drivers
Description: Size of drivers ablated
Time Frame: Baseline
Population: Participant screen failed
Arm/Group | Patients With Atrial Fibrillation (AF)
Number analyzed (Participants) | 0

4. Secondary Outcome: Percent Change of Driver Regions
Description: Percent change of driver regions after ibutilide
Time Frame: Baseline and 1 year
Population: Participant screen failed
Arm/Group | Patients With Atrial Fibrillation (AF)
Number analyzed (Participants) | 0

5. Secondary Outcome: AF Termination Rate
Description: AF termination rate is defined as AF termination to AT/SR (Atrial Tachycardia/Sinus Rhythm)
Time Frame: post ablation inducibility of AF after 5 minutes of burst pacing
Population: Participant screen failed
Arm/Group | Patients With Atrial Fibrillation (AF)
Number analyzed (Participants) | 0

6. Secondary Outcome: Total Procedure Time
Description: Total duration of RF ablation/fluoroscopy time/exposure procedure time
Time Frame: within 24 hours after the procedure is completed the time is calculated
Population: Participant screen failed
Arm/Group | Patients With Atrial Fibrillation (AF)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Participant screen failed
Arm/Group | Patients With Atrial Fibrillation (AF)
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT03370536/Prot_SAP_000.pdf